CLINICAL TRIAL: NCT04942392
Title: Digital Dance for People With Parkinson's Disease During the COVID-19 Pandemic: A Feasibility Study
Brief Title: Digital Dance for People With Parkinson's Disease During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Karlstad University (Other)
Responsible Party: Principal Investigator, Anna Stigsdotter Neely, Professor, Umeå University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 136/2019
Record Dates: First submitted 2021-06-23; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- digital dance for PD (Experimental)
  Interventions: Device: Digital dance for PD

INTERVENTIONS:
Device: Digital dance for PD — The digital dance class was held via Zoom. The class was scheduled once a week for 60 min and consisted of 10 sessions. A professional, certified Dance for PD and experienced dance instructor was teaching the dance class. The dance classes followed the Dance for PD protocol yet was adjusted to fit the digital zoom format.

SUMMARY:
Dance as a treatment to support physical, cognitive and emotional functioning, has gained increased acceptance as a healthcare intervention for people with Parkinson's Disease (PD). The impact of the COVID-19 pandemic has been far reaching with devastating effects for at-risk populations. To find alternative and safe treatment delivery options during the pandemic has been of outmost importance.

This mixed-methods, feasibility study on digital for people with Parkinson's Disease aimed to investigate: (1) the feasibility and safety of a digital home-based dance intervention for people with PD; (2) change in self-reported quality of life, cognitive complaints, psychological health and fatigue; and (3) the experience of digital dance for people with PD.

Twenty-three participants partook in 10 weekly digital dance classes at home via zoom. Feasibility outcomes measures were administered at post-test. Pre-post changes in self-reported quality of life, cognitive complaints, psychological health and fatigue were measured, as well as the experience of digital dance via focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported diagnosis of Parkinson's Disease
* Participant in Dance for PD at Balettakademien, Stockholm, Sweden

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome measures | Assessed at post-test
  The following feasibility outcome measures were assessed: (a) Technical and safety issues, (b) Compliance and motivation, (c) Self-assessed improvement in physical function, wellbeing and cognitive function and (d) The importance of dance as an artistic and creative activity.
  Each feasibility outcome measure was assessed via a 5-point Likert scale ranging from (1=very unsatisfactory, 5=very satisfactory), (1=not motivated, 5=very motivated), (1=noticeable worsening, 5=noticeable improvement) or (1=not meaningful, 5=very meaningful). Furthermore, each feasibility outcome measure had an open-ended question connected to it in order to capture any details related that feasibility domain. Two open-ended questions regarding positive and negative aspects of digital dancing were also included.
  For each feasibility outcome measure, a criterion of success was developed in order to judge the the success rate of these feasibility outcome measures.

SECONDARY OUTCOMES:
Depression and anxiety | 12 weeks (pretest - posttest)
  Severity of depression and anxiety symptoms measured by Hospital Anxiety Depression scale Anxiety score: 0-21 higher score indicate more anxiety Depression score: 0-21 higher score indicate more depression
Quality of life (QoL) Summary index | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39), Summary index: 0-100 higher scores indicate more problems.
  Furthermore, scores on the following subscales were assessed:
  * Mobility score: 0-100 higher scores indicate more problems
  * Activity of Daily Living score: 0-100 higher scores indicate more problems
  * Emotional well being score: 0-100 higher scores indicate more problems
  * Stigma score: 0-100 higher scores indicate more problems
  * Social support score: 0-100 higher scores indicate more problems
  * Cognition score: 0-100 higher scores indicate more problems
  * Communication score: 0-100 higher scores indicate more problems
  * Bodily discomfort score: 0-100 higher scores indicate more problems
Quality of life (QoL) - Bodily discomfort | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale: Bodily discomfort score: 0-100 higher scores indicate more problems
Quality of life (QoL) Communication | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale: Communication score: 0-100 higher scores indicate more problems
Quality of life (QoL) Cognition | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale:Cognition score: 0-100 higher scores indicate more problems
Quality of life (QoL) Social support | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale: Social support score: 0-100 higher scores indicate more problems
Quality of life (QoL) Stigma | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale: Stigma score: 0-100 higher scores indicate more problems
Quality of life (QoL) Emotional well being | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale: Emotional well being score: 0-100 higher scores indicate more problems
Quality of life (QoL) Activity of Daily Living | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale: Activity of Daily Living score: 0-100 higher scores indicate more problems
Quality of life (QoL) - Mobility | 12 weeks (pretest - posttest)
  Quality of life measured by Parkinson's Disease Questionnaire-39 (PDQ39).
  Subscale Mobility score: 0-100 higher scores indicate more problems
Fatigue | 12 weeks (pretest - posttest)
  Fatigue measured by Checklist Individual Strength Questionnaire (CIS). Total score: 20-140
Subjective cognitive complaints | 12 weeks (pretest - posttest)
  Improvement on subjective memory complaints measured by Prospective Retrospective Memory Questionnaire (PRMQ). Total score: 16-80 higher scores indicate more cognitive complaints prospective score: 0-100 higher scores indicate more cognitive complaints retrospective score: 0-100 higher scores indicate more cognitive complaints short term score: 0-100 higher scores indicate more cognitive complaints long term score: 0-100 higher scores indicate more cognitive complaints self cued score: 0-100 higher scores indicate more cognitive complaints environmentally cued: 0-100 higher scores indicate more cognitive complaints
Mental fatigue | 12 weeks (pretest - posttest)
  Two questions from the Mental Fatigue Scale were used to measure mental fatigue (item 3) and recovery (item 4). Answers were given on a 7-point Likert scale.
Experience and meaning of digital dance for people with PD | Assessed at post-test
  Two focus group interviews were conducted to examine the broader experience of digital dance for people with PD.

OTHER OUTCOMES:
Age | Assessed at pre-test
  Demographic characteristic: age at baseline
Sex | Assessed at pre-test
  Demographic characteristic: sex
Educational level | Assessed at pre-test
  Demographic characteristic: educational level
Previous experience of dance for Parkinson's Disease | Assessed at pre-test
  Demographic characteristic: previous experience of dance for PD
Self-evaluated health | Assessed a pre-test
  Demographic characteristic: self-evaluated health
Disease duration | Assessed at pre-test
  Demographic characteristic: self-reported year of PD diagnosis
Current participation in physical exercise | Assessed at pre-test
  Demographic characteristic: current participation in physical exercise

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Neely, prof, Principal Investigator — Umeå University
Locations (1):
- Balettakademien, Stockholm, Sweden

REFERENCES:
- [Derived] Walton L, Domellof ME, Astrom AN, Elowson A, Neely AS. Digital Dance for People With Parkinson's Disease During the COVID-19 Pandemic: A Feasibility Study. Front Neurol. 2022 Feb 3;12:743432. doi: 10.3389/fneur.2021.743432. eCollection 2021. PMID 35185746